CLINICAL TRIAL: NCT06846736
Title: ALK Digital Pathology Outcome Prediction
Brief Title: ALK Digital Pathology Outcome Predition, Multi Institutional, Restrospective Study
Acronym: ALKDigPath
Status: Enrolling by invitation | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Mayo Clinic (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Other Study IDs: SMC-9969-22
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-08

CONDITIONS: Alk-positive Non-Small Cell Lung Cancer; ALK-inhibitor Treated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Goal of this observational study is to develop an AI-driven pathologic image analysis-based classifier that can identify patients unlikely to significantly benefit from the currently utilized first-line ALK inhibitors (advanced-generation ALK inhibitors). Our goal is a classifier with final ROC-AUC value of 0.75.

DETAILED DESCRIPTION:
This is a retrospective study. All data have been collected at different time points during the patients' routine visits at the hospital.

1. Collection of a retrospective set of ALK positive patients with advanced NSCLC that have received an advanced-generation ALK inhibitor treatment as the first ALK inhibitor (i.e. alectinib, lorlatinib, brigatinib or ceritinib): collection of the clinical data, pathologic data, response to treatment and scans H&E images
2. Image analysis of the scanned H&E images, development of a classifier of the data to identify responders vs. non-responders.

Image analysis and AI development will be carried out at the Sheba Medical Center, in-house development. The clinical data will be analyzed, tagging study samples as belonging to a responder (R), vs. a non-responder (NR). For the purpose of this study, a NR will be defined as a patient that has progressed or died on an ALK inhibitor treatment within the first year of treatment.

The study cases will be randomly split to three: a training cohort, a validation cohort and a test cohort. The cohorts will be stratified by the response to treatment (i.e. equal proportion of R vs. NR cases in each cohort). Next, scanned images will be processed and analyzed. Slides analysis would be done using python using the pytorch packages. Further statistical analysis will be done with R statistical programming.

At first the whole slide image (WSI) is divided into thousands of tiles. These are examined by a convolutional neural network (CNN) to extract tile level features. We will be using Resnet, a common deep learning model used for computer vision as the CNN. The CNN will be trained with multiple instance learning (MIL) at the tile level and later the predicted scores will be aggregated for the WSI level . The final model will be conducted on the slides, to distinguish between R vs. NR. The classifier will be developed on the training cohort, modified if required following processing of the validation cohort and finally tested for efficacy on the test cohort. Cross-Validations techniques will also be used.

We aim to use this technique in order identify a sub-group of ALK positive patients that might be candidates for more aggressive treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years;
* Patient with an oncologic disease;
* ALK positive patients with advanced NSCLC that have received an advanced-generation ALK inhibitor treatment as the first ALK inhibitor (i.e. alectinib, lorlatinib, brigatinib or ceritinib)

Exclusion Criteria:

* Absence of information on the last oncologic treatment received;
* Patient without a general or specific consent for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALK positive patients with advanced NSCLC that have received an advanced-generation ALK inhibitor treatment as the first ALK inhibitor
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-08-13 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
A classifier predicting outcome for advanced NSCLC ALK+ patients on ALK inhibitor treatment | 36 months
  A classifier predicting outcome for advanced NSCLC ALK+ patients on ALK inhibitor treatment, based on AI analysis of digital pathology images of the diagnostic biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Jair Bar, MD-PhD, Principal Investigator — Sheba Medical Cernter
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Based on inidividual requests

DOCUMENTS (1):
  • Study Protocol (2024-09-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT06846736/Prot_000.pdf